CLINICAL TRIAL: NCT05885178
Title: Triage of Patients With Acute Ischemic Stroke Due to Large Vessel Occlusions-1 (TRACK-LVO-1): an Imaging-based Patient Registry Study
Brief Title: Triage of Patients With Acute Ischemic Stroke Due to Large Vessel Occlusions-1 (TRACK-LVO-1)
Acronym: TRACK-LVO-1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Other Study IDs: TJHH-2023-WeiMing
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute Ischemic; Endovascular Procedures; Large Vessel Occlusion
Keywords: Acute Ischemic Stroke; Endovascular Therapy; Large Vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Endovascular therapy: Timely thrombectomy for acute ischemic stroke patients with large vessel occlusion by either stent retriever, thrombus aspiration, others, or combination methods.
  Interventions: Procedure: Endovascular Therapy
- Best medical management: Patients enrolled in this group received the best medical management.
  Interventions: Procedure: Endovascular Therapy

INTERVENTIONS:
Procedure: Endovascular Therapy — Endovascular therapy, as an adjunct to standard stroke therapy, may be beneficial for a very select population of patients who present with an acute ischemic stroke and have a proven large, proximal occlusion on imaging.
  Endovascular therapy includes any one or more of the following:
  Intra-arterial thrombolytic therapy, aspiration, stent retrieval, or a combination of multiple mechanical devices.

SUMMARY:
The aim of this study is to establish an academic, real-world, single-center, observational registry of consecutive patients hospitalized with acute ischemic stroke (AIS) due to large vessel occlusions (LVO), treated with either endovascular therapy (EVT) or best medical management (BMM).

DETAILED DESCRIPTION:
Stroke is a major threat to public health and is exacerbating socioeconomic development. It is the leading cause of mortality among residents in China. Large vessel occlusion (LVO) is a predictor of unfavorable outcomes and can account for up to 52% of patients with acute ischemic stroke (AIS). The definition of LVO and its optimal screening imaging modalities remain controversial. In this registry, the investigators defined LVO as an occlusion of the intracranial ICA with or without the involvement of the terminal bifurcation, M1 and/or M2 segment of the MCA, A1 and/or A2 segment of the ACA, VA, BA, or P1 and/or P2 segment of the PCA.

TRACK-LVO is an academic, real-world, single-center, observational registry, in which consecutive patients hospitalized with AIS due to LVO will be treated with either EVT or BMM. Baseline information and clinical follow-up information at 90 days from stroke onset are collected. The key baseline items in this registration for both EVT and BMM groups include basic demographic profiles, past medical history, NIHSS score, treatment with intravenous alteplase, type of stroke onset, time from stroke onset to admission/imaging, imaging characteristics such as the volume of the ischemic core and occlusion site, and treatment-related complications. Additional information collected in EVT groups includes details of EVT procedure and angiographic images.

The investigators enrolled patients with LVO screened under different imaging modalities to further reveal the optimal imaging modalities in the detection of LVO. The investigators also tend to compare the prognosis of AIS patients with LVO receiving endovascular therapy and the best medical management respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patient admitted from Jan. 1st, 2018 to June. 1st, 2021;
2. Age ≥ 18;
3. Ischemic stroke confirmed by head CT or MRI;
4. Large vessel occlusion confirmed by head CTA or MRA: intracranial internal carotid artery (ICA), middle cerebral artery (MCA M1/M2), anterior cerebral artery (ACA A1/A2), basilar artery (BA), vertebral artery (VA), and posterior cerebral artery (PCA P1/P2);
5. Patients receiving either endovascular therapy or best medical treatment;

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke due to large vessel occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Modified ranking scale (mRS) at 90 days | 90 days
  A 0-6 scale running from perfect health without symptoms to death.
Mortality within 90 days | 90 days
  mortality of any causes.

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) scores at 90 days | 90 days
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Occurrence of periprocedural complications | 14 days postoperatively
  Periprocedural complications include any intracranial hemorrhage, cerebral edema, brain herniation and pneumonia.
ASPECT score (Alberta Stroke Program Early CT score) | Day 0
  ASPECTS is a 10-point quantitative topographic CT scan score used in patients with middle cerebral artery (MCA) stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China